CLINICAL TRIAL: NCT04140591
Title: Proton Pump Inhibitor Plus Propranolol Versus Proton Pump Inhibitor Alone on Peptic Ulcer Healing in Patients With Liver Cirrhosis: a Randomized Trail
Brief Title: Proton Pump Inhibitor Plus Propranolol Versus Proton Pump Inhibitor Alone on Peptic Ulcer Healing in Patients With Liver Cirrhosis
Acronym: PU
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: 1. Most patients with liver cirrhosis already use PPI and NSBB 2. 90 % Peptic ulcer size is smaller than 5cm
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, The Division of Gastroenterology & Hepatology, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V106C-137
Record Dates: First submitted 2019-08-29; First posted 2019-10-28 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2019-09

CONDITIONS: Liver Cirrhosis; Peptic Ulcer
Keywords: Portal hypertension; Peptic ulcer; Non-selective beta-blocker; Proton pump inhibitor
MeSH Terms: conditions — Liver Cirrhosis; Peptic Ulcer; Hypertension, Portal | interventions — Proton Pump Inhibitors; Propranolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

ARMS (2):
- Proton-pump inhibitor (Placebo Comparator): PPI: Pariet EC 20 mg/QDAC
  Interventions: Drug: Proton-pump inhibitor
- Propranolol+Proton-pump inhibitor (Active Comparator): Propranolol:
  Propranolol 10mg BID initially and titrate dosage every week to achieve 25% drop of heart rate (keep heart rate>55 or systemic blood pressure>90mmHg)
  PPI: Pariet EC 20 mg/QDAC
  Interventions: Drug: Propranolol+Proton-pump inhibitor

INTERVENTIONS:
Drug: Proton-pump inhibitor — PPI: Pariet EC 20mg/QDAC
  Other Names: Pariet EC; PPI
  Arms: Proton-pump inhibitor
Drug: Propranolol+Proton-pump inhibitor — Propranolol 10mg BID initially and titrate dosage every week to achieve 25% drop of heart rate (keep heart rate>55 or systemic blood pressure >90mmHg) PPI: Pariet EC 20mg/QDAC
  Other Names: Inderal; Cardolol
  Arms: Propranolol+Proton-pump inhibitor

SUMMARY:
Proton pump inhibitor plus propranolol versus proton pump inhibitor alone on peptic ulcer healing in patients with liver cirrhosis: a randomized trail

DETAILED DESCRIPTION:
Portal hypertension is responsible for the development of portosystemic collaterals. The hemodynamic alternations may result in mucosal and vascular changes along gastrointestinal (GI) tract as well. According to several epidemiological studies, cirrhotic patients are at a higher risk of developing peptic ulcers, delayed healing, and a higher frequency of ulcer recurrence. The death rate from peptic ulcer disease in cirrhotic patients has been reported to be five times higher than that of the general population. The exact mechanism remains incompletely understood, but may be related to impaired mucosal defense mechanisms. Aggressive factors such as Helicobacter pylori and gastric acid may not be the predominant etiology in such circumstances. Sarfeh et al. found gastric mucosa of portal hypertensive rats, compared with that of controls, has distinctive functional and histologic abnormalities that can explain its increased susceptibility to erosive injury. Auroux et al. found gastroduodenal ulcer was independently associated only with the severity of the hypertensive gastropathy in cirrhotics. Chen et al. found portal hypertension with a hepatic venous pressure gradient > 12 mmHg may be an important factor contributing to the increased prevalence of gastric ulcer observed in patients with liver cirrhosis. Thereby, we presumed that clinically significant portal hypertension may play a role in development of peptic ulcer in cirrhotic patients. Lebrec et al. elucidated non-selective beta-blocker (NSBB) could significantly decrease portal pressure and lower the risk of GI bleeding in patients with cirrhosis. Kitano et al. found portal hypotensive treatment with NSBB, reduces ethanol-induced gastric mucosal damage in portal hypertensive rats and improves endoscopic signs of portal hypertensive gastropathy in cirrhosis patients. We designed a 2-year randomized trial to evaluate the effectiveness of proton pump inhibitor with or without propranolol on ulcer healing and the incidence of ulcer bleeding in patients with cirrhosis and peptic ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 and 85 years old
* Liver cirrhosis associated with esophageal varices or gastric varices
* Gastric ulcer or duodenal ulcer ,size bigger or egual than 0.5 cm

Exclusion Criteria:

* Acute bleeding
* Steroid or NSAID user
* Pregnancy, or the patients with other terminal illness (such as other terminal cancers, heart failure, renal failure...)
* Propranolol contraindications (such as atrioventricular block, heart failure, chronic obstructive pulmonary disease, asthma, poorly controlled diabetes, severe peripheral arterial disease...)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12-26 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Healing of peptic ulcer | 2 months
  if propranolol can help cure peptic ulcer
Bleeding rate of peptic ulcer | 2 months
  if propranolol can help decrease the rate of ulcer bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chih mchou@vghtpe.gov.tw, MD, Principal Investigator — Institutional Review Board, Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taiwan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided